CLINICAL TRIAL: NCT04423653
Title: The Feasibility and Trend of Functional Changes by Using Home-based Exercise Program Delivered Through Telehealth With Coaching for Adolescents With Spastic Cerebral Palsy
Brief Title: The Feasibility of Telehealth HEP for CP (HEP: Home Exercise Program), (CP: Cerebral Palsy)
Acronym: HEPCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00145690
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Cerebral Palsy, Spastic; Telemedicine
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-coaching group (Experimental): This group will receive exercises videos, 2 sessions a week to be done on participant's own and the 3rd session will be live video conference session for training, supervision, and consultation purposes.
  Interventions: Behavioral: Telehealth home exercise program
- Self-monitored group (Active Comparator): This group will receive exercises videos, 3 sessions a week to be done on participant's own with out any supervision.
  Interventions: Behavioral: Telehealth home exercise program

INTERVENTIONS:
Behavioral: Telehealth home exercise program — The intervention will include videos of exercises and also live coaching using telehealth system.

SUMMARY:
This study will provide exercise videos and live consultation sessions for adolescents with spastic cerebral palsy. We will recruit 20 participants with 10-18 years old and will be randomized into an experimental or control group. The experimental group will receive exercises videos 2 times a week and one time live consultation session for 8 weeks.

The Control group will receive exercise videos 3 times a week for 8 weeks. Both groups will use HIPAA compliant telehealth provider (Physitrack website/ app).

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with spastic CP diagnosis, Gross Motor Functional Classification System (GMFCS) levels I-III) which will be confirmed by GMFCS-Extended Revised.
* Between the ages of 11 and 18 years old.
* Having a stable health status for 6 weeks prior to screening.
* Having the cognitive ability to follow an exercise instruction in either written or electronic format, with or without support from their parents.
* With an approval from parents/guardians for participating in this study.
* Having access to the internet at home and access to the exercise's website/app via Personal computer (PC), laptop, or mobile app.
* Being able to understand and follow verbal commands in English. The intervention and the questionnaires are available in English only.

Exclusion Criteria:

Subjects will be excluded if they have:

* unstable medical condition during past 6 weeks,
* had other neurological disorders that may cause further decline in balance and walking abilities (head injury, vestibular dysfunction, or Spinal cord injury),
* or any musculoskeletal condition that would interfere with the safe performance of the exercise intervention or testing protocol,
* scheduled surgical operations or castings during study period,
* scheduled for intensive rehabilitation during 8 weeks of intervention.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | post-intervention (after end of 8-weeks)
  Recruitment rate will be calculated as the total number of patients recruited, divided by the maximum number of sites and then divided by the average number of months recruiting
Adherence Rate | post-intervention (after end of 8-weeks)
  Adherence will be calculated as numbers: practice days, sessions, exercises, and repetitions.
Compliance Rate | post-intervention (after end of 8-weeks)
  Compliance rate will be calculated by number of participants who will complete the whole intervention duration and be examined post-intervention.
Canadian occupational performance measure score change | Baseline, Post-intervention (after end of 8-weeks)
  Achievements of individualized goals will be measured using the adapted version of COPM.
  For our study, 1-3 individualized goals are determined together by the parents/guardians, physical therapist, and investigators during the 2nd baseline visit. Children/parents will rate the current level of performance of each goal on scale 1-10 and satisfaction level of performance on scale 1-10, during the videoconferencing session along with physical therapist and investigators. The change in scores will be calculated (post-intervention score - Baseline score)

SECONDARY OUTCOMES:
The physical activity questionnaire for children (PAQ-C) and for Adolescents (PAQ-A) | Baseline, Post-intervention (after end of 8-weeks)
  The physical activity questionnaire for children (PAQ-C) and for Adolescents (PAQ-A) versions will be used to evaluate Physical activity level. The PAQ is self-administered, 7-day recall instrument. It is to assess general levels of physical activity in school students between 8-19. PAQ-C has 9 items while PAQ-A has 8 items, and each item is ranked on a 5-point scale. Both versions showed validity and reliability.
The Physical Activity and Enjoyment Scale (PACES) | Baseline, Post-intervention (after end of 8-weeks)
  This questionnaire consists of 16 statements that are scored on a five-point rating scale (1 = disagree a lot, 5 = agree a lot).
The Cerebral Palsy Quality of Life Questionnaire (CP-QOL) | Baseline, Post-intervention (after end of 8-weeks)
  The Cerebral Palsy Quality of Life Questionnaire for Children (CP QOL-Child) and Cerebral Palsy Quality of Life Questionnaire for Adolescents (CP QOL-Teen) will be utilized to evaluate the QOL either using the self-reported version or proxy-parent report.
  The CP QOL-Child is to assess the quality of life of children with cerebral palsy aged 4-12 years. An adolescent version, the CP QOL-Teen, has recently been developed for adolescents aged 13-18 years. It assesses different domains including social wellbeing & acceptance, Feelings about functioning, Participation & physical health, Emotional wellbeing & self-esteem, Access to services, Pain & impact of disability, Family health.
The Correctness of Exercise Performance (COEP) | Baseline, halfway of intervention (after end of 4-weeks), Post-intervention (after end of 8-weeks)
  (COEP) scale will be used to grade the quality of performance based on three criteria: 1) the performance has been carried out so well that the goal of the exercise is reached, 2) the exercise is not performed correctly and the goal is not reached, although no negative effect is to be expected, and 3) the exercise is carried out incorrectly, the goal is not reached and there is reason to assume that the exercise causes harm. Participants will be videotaped while they are performing the prescribed exercises at home, by parents and videos will be shared with investigator.
Telehealth Usability Questionnaire (TUQ) | Post-intervention (after end of 8-weeks)
  TUQ is 21 questions with a score ranging from 1 to 7 for each question.
pediatric pain questionnaire (PPQ) | Baseline, Post-intervention (after end of 8-weeks)
  To assess pain intensity and location and the sensory, affective, and evaluative qualities of pain, appropriate for children and adolescents. Visual Analogue scale (VAS) describing pain intensity, body outline to describe location of pain, and words describing pain to assess qualities of pain.
Children Sleep Habits Questionnaire(CSHQ) | Baseline, Post-intervention (after end of 8-weeks)
  is a 45-item, parent-rated questionnaire that assesses the frequency of behaviors associated with common pediatric sleep difficulties.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Will share only aggregate and overall project results through poster and/or oral presentations at local, regional and national meetings.

REFERENCES:
- [Background] Buffart LM, Westendorp T, van den Berg-Emons RJ, Stam HJ, Roebroeck ME. Perceived barriers to and facilitators of physical activity in young adults with childhood-onset physical disabilities. J Rehabil Med. 2009 Nov;41(11):881-5. doi: 10.2340/16501977-0420. PMID 19841838
- [Background] Lai B, Young HJ, Bickel CS, Motl RW, Rimmer JH. Current Trends in Exercise Intervention Research, Technology, and Behavioral Change Strategies for People With Disabilities: A Scoping Review. Am J Phys Med Rehabil. 2017 Oct;96(10):748-761. doi: 10.1097/PHM.0000000000000743. PMID 28398967
- [Background] Fauzi AA, Khayat MM, Sabirin S, Haron N, Mohamed MNA, Davis GM. Structured home-based exercise program for improving walking ability in ambulant children with cerebral palsy. J Pediatr Rehabil Med. 2019;12(2):161-169. doi: 10.3233/PRM-180538. PMID 31227664
- [Background] Novak I, Berry J. Home program intervention effectiveness evidence. Phys Occup Ther Pediatr. 2014 Nov;34(4):384-9. doi: 10.3109/01942638.2014.964020. Epub 2014 Oct 15. No abstract available. PMID 25317927
- [Background] Novak I. Effective home programme intervention for adults: a systematic review. Clin Rehabil. 2011 Dec;25(12):1066-85. doi: 10.1177/0269215511410727. Epub 2011 Aug 10. PMID 21831927